CLINICAL TRIAL: NCT05835076
Title: Helicobacter Pylori Screening in Hyperemesis Gravidarum in Early Pregnancy
Brief Title: Helicobacter Pylori Screening at Sohag University
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Amr Ayman Hassan, Helicobacter pylori screening in hyperemesis gravidarum in early pregnancy, Sohag University
Other Study IDs: Soh-Med-23-04-03MS
Record Dates: First submitted 2023-04-18; First posted 2023-04-28 (Actual); Last update posted 2023-04-28 (Actual); Status verified 2023-04

CONDITIONS: In Early Pregnancy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Stool antigen test — Antigen test in the stool analysis

SUMMARY:
Screen of Helicobacter pylori in hyperemesis gravidarum in early pregnancy to detect the impact of the severity of the disease on pregnant women

ELIGIBILITY:
Inclusion Criteria:

* pregnant woman <16wk

Exclusion Criteria:

* pregnant woman >16wks

Ages: 18 Years to 40 Years | Sex: Female
Age Groups: Adult
Gender Based: Yes — Pregnant women
Study Population: Cross sectional study to screen Helicobacter pylori in hyperemesis gravidarum
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2023-04 (Estimated); Primary Completion 2024-04 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Positive | 2 days
  Positive for Helicobacter pylori

IPD SHARING:
Plan to Share IPD: Undecided